CLINICAL TRIAL: NCT00032864
Title: Clinical Trial of Footwear in Patients With Diabetes
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: S003
Record Dates: First submitted 2002-04-04; First posted 2002-04-05 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2003-02

CONDITIONS: Amputations; Diabetes; Lower Extremity Ulcers
Keywords: amputations, diabetes,
MeSH Terms: conditions — Diabetes Mellitus; Leg Ulcer

SUMMARY:
A Seattle VA study indicated lower extremity ulcers preceded 84% of diabetic amputations. Nearly half of the events that ban the causal chain leading to ulcers and amputation were initiated by ill-fitting footwear. Other investigators report similar findings for injurious footwear in their diabetic patient populations. Yet, the efficacy of footwear in preventing ulcers and amputations in the high-risk diabetic population has received limited experimental investigation. A British descriptive study followed diabetic patients with healed foot ulcers for two years and found reulceration occurred in 72% of patients who resume wearing their own footwear compared to 26% of patients who continued wearing "prescribed" footwear. A Swedish cohort study identified individuals with a foot ulcer and reported their 1, 3, and 5 year reulceration rates at 34%, 61%, and 70%, respectively, without further specifying footwear components. In a German diabetic population the reulceration rate was 87% in-patients who abandoned their custom shoes and resumed wearing their own shoes compared to 42% of those who continued to wear their custom shoes. Unfortunately, none of these studies compared the single or combined contribution of therapeutic shoes or insoles on foot ulcer prevention. Nor did these studies address patient adherence to prescribed footwear; thus the actual efficacy of various footwear interventions in foot ulcer prevention in this high-risk population is still to be tested.

DETAILED DESCRIPTION:
Primary Objective:

Half of the 7,646 amputations performed in VA in 1996 were in veterans with diabetes. Lower extremity ulcers preceded about 85% of diabetic amputations. Minor trauma, often footwear or repetitive pressure related, initiated the majority of the ulcers. Persons with diabetes have unique footwear needs. In 1997, Gayle E. Reiber MPH, PhD, and Douglas G. Smith, MD of the VA Puget Sound Health Care System initiated a randomized clinical trial (1) to determine the extent to which study shoes and study inserts would reduce the incidence of re-ulceration in diabetic individuals with a prior foot ulcer history, and (2) to estimate costs of ulcer prevention using these strategies. A total of 400 patients from the VA Puget Sound Health Care System (n=189) and a Seattle-area Health Maintenance Organization, Group Health Cooperative (n=211), have now been randomized to one of three study arms: Arm 1 (n=120) study shoes and customized cork inserts; Arm 2 (n=119) study shoes and generic polyurethane inserts; and Arm 3 (n=161) controls who are wearing their own footwear. Patients in Arms 1 and 2 received formal, leisure and athletic shoes built to study specifications by Cole-Haan for men and by Lowell Shoe for women. Patients will be followed for two years to determine the incidence and cost of foot re-ulceration.

Study Abstract:

A Seattle VA study indicated lower extremity ulcers preceded 84% of diabetic amputations. Nearly half of the events that ban the causal chain leading to ulcers and amputation were initiated by ill-fitting footwear. Other investigators report similar findings for injurious footwear in their diabetic patient populations. Yet, the efficacy of footwear in preventing ulcers and amputations in the high-risk diabetic population has received limited experimental investigation. A British descriptive study followed diabetic patients with healed foot ulcers for two years and found reulceration occurred in 72% of patients who resume wearing their own footwear compared to 26% of patients who continued wearing "prescribed" footwear. A Swedish cohort study identified individuals with a foot ulcer and reported their 1, 3, and 5 year reulceration rates at 34%, 61%, and 70%, respectively, without further specifying footwear components. In a German diabetic population the reulceration rate was 87% in-patients who abandoned their custom shoes and resumed wearing their own shoes compared to 42% of those who continued to wear their custom shoes. Unfortunately, none of these studies compared the single or combined contribution of therapeutic shoes or insoles on foot ulcer prevention. Nor did these studies address patient adherence to prescribed footwear; thus the actual efficacy of various footwear interventions in foot ulcer prevention in this high-risk population is still to be tested.

Age Groups: Child, Adult, Older Adult
Dates: Start 1997-01; Study Completion 2000-09